CLINICAL TRIAL: NCT04062435
Title: Corneal Uptake of Riboflavin Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Katja Iselin, Principal Investigator, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCI_02
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Keratoconus
Keywords: Cross-linking, Riboflavin, Fluorophotometry, FluorotronTM Master
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Experimental): Peschke®TE 0.25 % application in the INFERIOR FORNIX
  Peschke®TE 0.25 % (Peschke Trade, Hünenberg, Switzerland) eye drops, 1 drop every 5 minutes over 60 minutes by the Principal Investigator.
  Interventions: Drug: Drop application in the inferior fornix
- Control Group (Active Comparator): Peschke®TE 0.25 % application on the CORNEA
  Peschke®TE 0.25 % (Peschke Trade, Hünenberg, Switzerland) eye drops, 1 drop every 5 minutes over 60 minutes by the Principal Investigator.
  Interventions: Drug: Drop application on the cornea

INTERVENTIONS:
Drug: Drop application in the inferior fornix — See Arms
  Arms: Interventional Group
Drug: Drop application on the cornea — See Arms
  Arms: Control Group

SUMMARY:
The overall objective of this study is to optimise the corneal cross-linking standard protocol in terms of a more economical use of the resource "medical personnel" and in terms of increased patient participation. If it can be shown that the riboflavin necessary for corneal cross-linking does not necessarily have to be applied directly on the cornea (as currently performed by the nurses), but can also be applied in the inferior fornix (as it would be performed by patients in the context of self-application), then it would be conceivable to transfer this task from medical staff to the patients.

DETAILED DESCRIPTION:
This national single-centre, experimental, randomized and controlled trial will comprise two parallel arms. The intervention to be studied will be an alternative application of riboflavin drops in the inferior fornix. As comparator serves a conventional riboflavin drop application directly on the center of the cornea. Our research hypothesis is that the application of riboflavin drops in the inferior fornix is not inferior to the corneal application with respect to the resulting riboflavin concentrations in the anterior chamber; which represents a sufficient corneal impregnation with riboflavin. This study is randomized but not blinded. Recruitment is anticipated to start in September 2019 and is scheduled to last 1-2 months. We will enroll 12 patients in each trial arm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy clinical staff members of the Dept. of Ophthalmology at the Lucerne Cantonal Hospital will be evaluated for study inclusion.
* Signed written informed consent form

Exclusion Criteria:

* Aged < 18 years
* Any ocular or systemic diseases with ocular side effects
* Medication with potential ocular side effects
* Epilepsia, due to the flickering light of the fluorophotometer used to measure anterior chamber riboflavin concentration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Quantitative changes in anterior chamber riboflavin concentrations over a time period of 60 min for both application sites (inferior fornix and cornea) | Three hours
  Correlating to our standard CXL protocol, the application phase lasts 60 min and the riboflavin drops will be applied by the principle investigator every 5 minutes on the cornea in the conventional and in the inferior fornix in the interventional group. The drop application will be performed in an upright position and without an eyelid speculum. During the application phase, fluorophotometric measurements will be repeated every 15 minutes and changes in corneal and anterior chamber riboflavin concentrations will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Iselin, MD, Principal Investigator — Dept. of Ophthalmology, Lucerne Cantonal Hospital
Locations (1):
- Dept. of Ophthalmology, Lucerne Cantonal Hospital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No